CLINICAL TRIAL: NCT01485302
Title: A Multi-center, Parallel-group, Double-blind, Placebo-controlled Single and Multiple Dose Escalation Study to Assess the Safety and Tolerability and the Pharmacokinetic Properties of SAR228810 Given as IV Infusion or as SC Injection in Patients With Mild to Moderate Alzheimer's Disease.
Brief Title: Single and Repeated Dosing Study to Assess the Safety and the Concentration-time Profile of SAR228810 in Alzheimer's Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDR12399; 2011-002910-35 (EudraCT Number); U1111-1120-0550 (Other: UTN)
Record Dates: First submitted 2011-11-16; First posted 2011-12-05 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Alzheimer's Disease
Keywords: mild to moderate Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): Dose 1 IV infusion
  Interventions: Drug: SAR228810
- Cohort 2 (Experimental): Dose 2 IV infusion
  Interventions: Drug: SAR228810
- Cohort 3 (Experimental): Dose 3 IV infusion
  Interventions: Drug: SAR228810
- Cohort 4 (Experimental): Dose 4 IV infusion
  Interventions: Drug: SAR228810
- Cohort 5 (Experimental): Dose 1 SC injection
  Interventions: Drug: SAR228810
- Cohort 6 (Experimental): Dose 2 SC injection
  Interventions: Drug: SAR228810

INTERVENTIONS:
Drug: SAR228810 — Pharmaceutical form:solution
  Route of administration: intravenous
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: SAR228810 — Pharmaceutical form:solution
  Route of administration: subcutaneous
  Arms: Cohort 5; Cohort 6

SUMMARY:
Primary Objective:

- To assess the safety and tolerability of escalating single and multiple doses of SAR228810 in patients with Alzheimer's disease (AD)

Secondary Objective:

- To evaluate the pharmacokinetic properties of SAR228810 after escalating single and multiple doses of SAR228810 in AD patients

DETAILED DESCRIPTION:
14.5 to 22 months

ELIGIBILITY:
Inclusion criteria:

* Male or female patients with mild to moderate Alzheimer's disease, aged between 50 and 85 years inclusive
* Meets criteria for probable Alzheimer's of the National Institute of Neurologic and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorders Association
* Mini-mental state examination (MMSE)
* In reasonable and stable health state for Alzheimer's patients of this age and stage of disease as assessed by a comprehensive clinical assessment
* Magnetic resonance imaging consistent with Alzheimer's disease, not indicating any other cause for dementia symptoms than Alzheimer's disease
* Rosen Modified Hachinski Ischemic score
* If on symptomatic treatment for Alzheimer's disease (acetylcholinesterase inhibitors or/and memantine), must be stable in the last 30 days before screening

Exclusion criteria:

* Clinically significant neurological disease other than Alzheimer's disease
* Had a major psychiatric disorder
* Had a history of stroke, seizures, brain neoplasms, brain surgery, or any cerebrovascular disorder (including transient ischemic attack)
* History or presence of severe, uncontrolled and/or unstable angiopathy or vasculitis.
* History or presence of clinically relevant cardiac disease.
* Currently taking anticonvulsants, anti-Parkinsonians, antipsychotics, anticoagulants or narcotic drugs, recent immunosuppressive or cancer chemotherapy drugs, or cognitive enhancers. Concomitant therapies that are allowed if given at a stable dose for at least 30 days before screening are: acetylcholinesterase inhibitors and/or memantine; antidepressants of the class of selective serotonin reuptake inhibitors (no tricyclics); acetyl salicylic acid (ASA) at a dose ≤ 160 mg/day;

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
number of patients with adverse events | 10 months

SECONDARY OUTCOMES:
AUC | 1 to 112 days after dosing
Cmax | 1 to 112 days after dosing
t1/2z | 1 to 112 days after dosing
brain magnetic resonance imaging | 10 months
hematology, biochemistry, coagulation | 10 months
vital signs, ECG | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- Investigational Site Number 100001, Sofia, Bulgaria
- France (2):
  - Investigational Site Number 250001, Pierre-Bénite
  - Investigational Site Number 250002, Toulouse
- Investigational Site Number 528001, Leiden, Netherlands
- Investigational Site Number 710001, Bloemfontein, South Africa
- Sweden (3):
  - Investigational Site Number 752003, Malmo
  - Investigational Site Number 752002, Mölndal
  - Investigational Site Number 752001, Stockholm